CLINICAL TRIAL: NCT05390021
Title: Diagnostic Performance of PET/MRI Versus Standard of Care Imaging (PET/CT and/or CT and/or PET) in Preoperative Women With Presumed Early-stage High Grade Endometrial Carcinoma
Brief Title: PET/MRI in Endometrial Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll patients to study
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Onofrio A. Catalano, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-112
Record Dates: First submitted 2022-05-18; First posted 2022-05-25 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Cytoreductive Surgery; Grade 3 Endometrial Endometrioid Adenocarcinoma; High Grade Serous Carcinoma; Endometrial Undifferentiated Carcinoma; Endometrial Mixed Cell Adenocarcinoma
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PET/MRI IN ENDOMETRIAL CANCER (Experimental): PET/MRI in one study visit of approximately four hours
  Interventions: Combination Product: PET/MRI with radiotracer ([18F]- fluorodeoxyglucose) and a gadolinium-based contrast agent

INTERVENTIONS:
Combination Product: PET/MRI with radiotracer ([18F]- fluorodeoxyglucose) and a gadolinium-based contrast agent — The research study procedures include a screening for eligibility and a single study visit. PET/MRI in one study visit of approximately four hours.

SUMMARY:
This study is investigating if positron emission tomography (PET)/Magnetic resonance imaging (MRI) is more effective than the currently used imaging modalities (computed tomography [CT], or PET/CT) for high-risk endometrial cancer.

The name of the intervention involved in this study is:

Positron Emission Tomography/Magnetic Resonance Imaging (PET/MRI)

DETAILED DESCRIPTION:
This research study involves undergoing a diagnostic imaging procedure called positron emission tomography/magnetic resonance imaging (PET/MRI). This type of scan uses a powerful magnet and a special drug that emits a small but detectable amount of radiation to show detailed images of tumors. This study, will examine the diagnostic effectiveness of positron emission tomography/magnetic resonance imaging (PET/MRI), which will be the intervention. The study will compare the results of this scan to either the computed tomography (CT) or PET/CT that participants would normally undergo as a standard of care for high-risk endometrial cancer.

The research study procedures include a screening for eligibility and a single study visit.

* Participants will undergo the PET/MRI in one study visit of approximately four hours.
* It is expected that about thirty-three (33) people will take part in this research study.

The U.S. Food and Drug Administration (FDA) has approved the PET/MRI scanner as a diagnostic modality option for indications that include for high-risk endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-85 years old with an endometrial biopsy-confirmed diagnosis of either grade 3 endometrioid, serous, carcinosarcoma, undifferentiated or mixed cell carcinoma
* Must have presumed stage I disease, i.e., no symptoms suggesting disease outside of the uterus (weight loss, early satiety, bloating, changes in bowel movement, etc.)
* Planning to undergo cytoreductive surgery with a Gynecologic oncologist employed by Massachusetts General Hospital
* No previous history of chronic severe renal insufficiency and a glomerular filtration rate of >30 mL/min/1.73m2. If the patient has a history of acute renal failure but their GFR as recovered to above 30,

Exclusion Criteria:

* Weight greater than 300lbs (the PET/MRI table weight limit) or BMI > 33
* Subjects less than 18 years of age or greater than 85 years of age
* Has Electrical implants, such as cardiac pacemakers or perfusion pumps
* Has Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, prosthetic heart valves that are not compatible with the gradient maps of our scanners, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, or steel implants not compatible with a 3 Tesla MR.
* Is actively anticipating being pregnant or breastfeeding (a negative STAT quantitative serum hCG pregnancy test is required on the day of the scan before the subject can participate)
* Suffers from claustrophobia
* If research-related radiation exposure exceeds current Radiology Department guidelines (i.e., 50 mSv in the prior 12 months)
* Is unable to lie comfortably on a bed inside the PET/MRI bore as assessed by physical examination and medical history (e.g., back pain, arthritis)
* Subject is under the direct professional supervision of the principal investigator
* A history of chronic severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73m2)
* Perioperative liver transplantation period

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a metastatic lesion noted on PET/MRI that have a true malignancy noted on surgical pathology of that lesion | Baseline
  Sensitivity of PET/MRI to detect metastatic lesions
Percentage of patients without any metastatic lesion noted on PET/MRI that do not have malignancy noted on surgical pathology | Baseline
  Specificity of PET/MRI to detect abscence of metastatic lesions

CONTACTS AND LOCATIONS:
Overall Officials: Onofrio Catalono, MD, PhD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation